CLINICAL TRIAL: NCT02601924
Title: Efficacy of Pressure Massage and Topical Gel on Pain During Inferior Alveolar Nerve Block and Maxillary Anterior Injections: A Single-Blind Randomized Clinical Trial
Brief Title: Efficacy of Pressure Massage and Topical Gel on Pain During Intra Oral Injections
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Nahid Mohammadzadeh Akhlaghi (Other)
Collaborators: Kerman University of Medical Sciences (Other)
Responsible Party: Sponsor-Investigator, Nahid Mohammadzadeh Akhlaghi, Associate Professor, Azad University of Medical Sciences
Organization: Azad University of Medical Sciences (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: KMU 1394.215
Record Dates: First submitted 2015-11-07; First posted 2015-11-11 (Estimated); Last update posted 2019-01-15 (Actual); Status verified 2019-01

CONDITIONS: Normal Pulp/ Pulpitis
Keywords: Anesthesia; injection; pain; pressure massage; topical gel
MeSH Terms: conditions — Pain

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Topical Pressure Massage Block injection (Active Comparator): Topical pressure massage at site of alveolar nerve block injection.
  Interventions: Other: Topical pressure massage
- Topical Anesthetic Gel Block injection (Active Comparator): Topical anesthetic gel (20% Benzocain) at site of inferior alveolar nerve block injection.
  Interventions: Drug: 20% Benzocain (Master-Dent, Monroe, NC)
- Topical Pressure Massage Infiltration (Active Comparator): Topical pressure massage at site of maxillary anterior infiltration
  Interventions: Other: Topical pressure massage
- Topical Anesthetic Gel Infiltration (Active Comparator): Topical anesthetic gel (20% Benzocain) at site of maxillary anterior infiltration
  Interventions: Drug: 20% Benzocain (Master-Dent, Monroe, NC)

INTERVENTIONS:
Drug: 20% Benzocain (Master-Dent, Monroe, NC) — Two topical anesthetic gel groups will receive anesthetic gel at the site of injection with massage on treating tooth.
  Other Names: Topical anesthetic gel
  Arms: Topical Anesthetic Gel Block injection; Topical Anesthetic Gel Infiltration
Other: Topical pressure massage — Two topical pressure massage groups will receive topical placebo gel with pressure massage at the site of injection.
  Arms: Topical Pressure Massage Block injection; Topical Pressure Massage Infiltration

SUMMARY:
Eighty patients with inclusion criteria will participate in this studyEach patient will receive an injection in one of the following groups according to the random number table:

1. Group TPMB: Topical pressure and massage with an Inferior alveolar nerve block (IANB)
2. Group TGB: Topical gel of 20% Benzocain (Master-Dent, Monroe, NC) with IANB
3. Group TPMI: Topical pressure and massage with a maxillary anterior infiltration (MAI)
4. Group TGI: Topical gel with a MAI. Immediately after the injection, patients will be asked to record the amount of pain they felt during needle penetration and injection using VAS form.Data will be analyzed using ANOVA and t-test.

DETAILED DESCRIPTION:
Eighty patients will be requested to take participate in this study after signing a written consent form. The inclusion criteria for the participants are as follows: 18-65 years old, having no systemic disease, not pregnant or beast feeding, having a mandibular premolar/molar or a maxillary anterior tooth with the diagnosis of normal pulp, reversible pulpitis or asymptomatic irreversible pulpitis (no or mild tenderness to percussion, normal periapical radiographic appearance), not taking analgesics, sedative or anti-anxiety medication and no intra oral injection at the treatment area, during the last 24 hours. By using a 170 mm Visual Analogue Scale (VAS), patients with pain less than or equal to 54 are classified as having asymptomatic irreversible pulpitis. The way to use the VAS will be explained to the patients prior to the procedure.

Each patient will receive an injection in one of the following groups according to the random number table:

1. Group TPMB: Topical pressure and massage with an Inferior alveolar nerve block (IANB)
2. Group TGB: Topical gel of 20% Benzocain (Master-Dent, Monroe, NC) with IANB
3. Group TPMI: Topical pressure and massage with a maxillary anterior infiltration (MAI)
4. Group TGI: Topical gel with a MAI

All the injections will be performed using an aspirating syringes containing 1.8 ml of lidocaine with 1:80000 epinephrine (2%Persocaine_E; Darupakhsh, Tehran, Iran) and 28-guage needles by a single operator (N.M.A). Immediately after the injection, patients will be asked to record the amount of pain they felt during needle penetration and injection using VAS form. If the patient is subjected to more than one injection during the root canal treatment, only the first injection will be subjected to the evaluation. Recording of the acquired data from the VAS forms will be done by another operator (P.M) who will be unaware of the patients' categorization.

Data will be analyzed using ANOVA and t-test with the significance level of p<0.05.

ELIGIBILITY:
Inclusion Criteria:

* Patients ranged18-65 years old
* No systemic disease
* Non pregnant or beast feeding
* A mandibular premolar/molar or a maxillary anterior tooth with the diagnosis of normal pulp, reversible pulpitis or asymptomatic irreversible pulpitis (Heft Parker visual analogue scale ≤ 54)
* Need dental treatment
* Not taking analgesics, sedative or anti-anxiety medication during the last 24 hours
* No intra oral injection at the treatment area during the last 24 hours

Exclusion Criteria:

-

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2016-02 (Actual); Primary Completion 2017-12 (Actual); Study Completion 2018-04 (Actual)

PRIMARY OUTCOMES:
Pain rate using Visual Analog Scale(VAS) | 2 minutes
  Topical anesthetic gel / pressure massage will be applied at the site of injection for 1 minute and anesthetic solution will be done during 1 minute